CLINICAL TRIAL: NCT06190288
Title: AdvantAGE: Implementation and Evaluation of an Interprofessional Transitional Care Model for Frail Older Adults at the University Department of Geriatric Medicine FELIX PLATTER
Brief Title: AdvantAGE: Implementation and Evaluation of an Interprofessional Tranistional Care Model for Frail Older Adults
Acronym: AdvantAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thekla Brunkert (Other)
Collaborators: Health Department of the Canton of Basel-Stadt (Other Government)
Responsible Party: Sponsor-Investigator, Thekla Brunkert, Principle Investigator, University Department of Geriatric Medicine FELIX PLATTER
Organization: University Department of Geriatric Medicine FELIX PLATTER (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 02072
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Transitional Care; Multimorbidity; Geriatric Care
Keywords: Transitional Care, Frailty, Rehospitalisation, Geratric Care
MeSH Terms: conditions — Frailty | interventions — imidacloprid

STUDY DESIGN:
Intervention Model Description: Hybrid effectiveness-implementation study (type 1)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The intervention includes five core elements provided by a multiprofessional team: (1) continuous support for patients and caregivers; (2) care coordination with primary care providers;(3) visits at patients' homes; (4) medication- and self-management with patients and caregivers; and (5) proactive advanced care planning. Patients will receive specialized support including home visits up to 90 days after hospital discharge.
  Interventions: Other: Transitional care model

INTERVENTIONS:
Other: Transitional care model — A newly developed care model to support frail older adults during their transition from hospital to home.
  Other Names: AdvantAGE

SUMMARY:
This clinical trial at the University Department of Geriatric Medicine FELIX Platter in Basel, Switzerland, is designed to evaluate a new transitional care model aimed at helping frail older adults after they get discharged from the hospital. The AdvantAGE study aims to explore the following questions:

* Does the new care model help reduce the number of patients who need to return to the hospital within 90 days?
* How effective is the implementation of this care model?

Participants in the trial will be followed by advanced practice nurses for up to 90 days after hospital discharge. The patients and their caregivers will receive support in coordinating care, managing medications, and learning to manage the patient's health conditions on their own. Additionally, they will have the opportunity to engage in discussions about advanced care planning.

ELIGIBILITY:
Inclusion Criteria:

* Currently admitted to the acute or rehabilitation ward of University Department of Geriatric Medicine
* Reside in Basel-Stadt
* Possess the ability to speak and comprehend the German language
* Scheduled to be discharged to their home
* 65 years or older
* Identified by a clinician as having a high risk of deterioration due to frailty

Additionally, participants must meet at least one of the following criteria:

* diagnosed with a complex chronic disease requiring support in self-management and disease management, or
* facing socially challenging situations such as living alone without a supportive network or lacking a GP, or
* admitted for an acute illness with a brief hospital stay (e.g., infection, cardiac decompensation) and need support in self- and disease management, and continuity of the therapy plan, including close monitoring.

Exclusion Criteria:

* residing in a nursing home or being newly admitted to one
* lacking informal caregivers and exhibiting severe cognitive impairment (MMS ≤23)
* scoring <50 on the motoric domain of the Functional Independence Measure (FIM)
* having a psychiatric disorder that significantly impacts their ability to manage daily life at time of the discharge

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
90-days rehospitalization rate | 90 days post-discharge
  Number of unplanned hospital admissions of any kind happening within 90 days after discharge

SECONDARY OUTCOMES:
30-days rehospitalization rate | 30 days post-discharge
  Number of unplanned hospital admission of any kind happening within 30 days after discharge
Time to readmission | Up to 90 days post-discharge
  Number of days between hospital discharge and unplanned hospital admission
Number of emergency room visits | 90 days post-discharge
  Number of emergency room visits (with or without hospital admission) within 90 days after discharge
Time to emergency room visit | Up to 90 days post-discharge
  Number of days between hospital discharge and emergency room visit
Patient's health-related quality of life | Up to 90 days post-discharge
  The EuroQoL-5D-5L is used to assess the health-related quality of life in patients at three time points. Prior to hospital discharge, 7 days and 90 days after hospital discharge or if the patient completed the intervention
Patient satisfaction questionnaire | up to 90 days post-discharge
  Satisfaction regarding intervention participation

CONTACTS AND LOCATIONS:
Overall Officials: Thekla Brunkert, PhD, Principal Investigator — Universitäre Altersmedizin FELIX PLATTER
Locations (1):
- Universitäre Altersmedizin FELIX PLATTER, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brunkert T, Pfundstein I, Nickel CH, Lampert ML, Trutschel D, Mauthner O. AdvantAGE: Implementation and Evaluation of an Interprofessional Transitional Care Model for Frail Older Adults-Protocol of an Effectiveness-Implementation Hybrid Study. J Adv Nurs. 2025 Aug;81(8):5130-5142. doi: 10.1111/jan.16745. Epub 2025 Jan 26. PMID 39865439
- See also: project homepage (in German) — https://advantage.nursing.unibas.ch/